CLINICAL TRIAL: NCT01128166
Title: Multisensor Chronic Evaluations in Ambulatory Heart Failure Patients
Brief Title: Evaluation of Multisensor Data in Heart Failure Patients With Implanted Devices
Acronym: MultiSENSE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MultiSENSE
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Decompensation; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients implanted with a CRT-D (Cardiac Resynch. Therapy)
  Interventions: Device: COGNIS CRT-D

INTERVENTIONS:
Device: COGNIS CRT-D — Patients with existing or newly implanted COGNIS® CRT-D pulse generators (PG)are enrolled in the study. PG is modified by the download of investigational software called Sensor Research Device-1™ (SRD-1). The goal of the SRD-1 system is to collect sensor data without affecting the delivered CRT-D therapy. This is accomplished through the "conversion" of an implanted COGNIS PG into a SRD-1 PG by downloading investigational software. Only a market approved COGNIS model N119/N120/P107/P108 device may be converted to a SRD-1 investigational device. There will be no PG hardware changes resulting from the conversion.

SUMMARY:
The goal of the MultiSENSE study is to collect chronic information from multiple sensors in an implanted device for evaluation in heart failure patients.

DETAILED DESCRIPTION:
The purpose of MultiSENSE study is to collect data about patient events during worsening heart failure, determine how sensor measurements vary during patient daily activities and during the development and recovery from events of worsening heart failure, develop algorithms capable of detecting the onset of worsening heart failure prior to the overt presentation of patient symptoms using reference measurements: thoracic impedance, heart sounds, physiologic responses to activities and respiration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of returning for all follow-up visits and emergency care at the investigational center as medically appropriate
* Willing to participate in all testing associated with this clinical investigation at an approved clinical investigational center
* Currently implanted with a COGNIS device (Model N119 or N120, P107, P108)
* Classified as NYHA Class II, III or IV within the last six months

Exclusion Criteria:

* Inability or refusal to sign the Subject Informed Consent
* Inability of refusal to comply with the follow-up schedule
* Documented as pacemaker dependent
* Unable to rest comfortably in a semi-recumbent position for up to 20 minutes
* Implanted with active Medtronic Fidelis lead models: 6930, 6931, 6948 or 6949
* Currently implanted with unipolar RA, RV, or LV leads
* LV sensitivity programmed to less than 0.7 mV AGC
* History of appropriate tachycardia therapy (external or implanted) for rates < 165 bpm within 1 week prior to enrollment
* Device battery status indicates approximate time to explant < 2 years
* Likely to undergo lead or PG revision during the course of the study as determined by the investigator
* Receiving regularly scheduled intravenous (IV) inotropic therapy as part of their drug regimen
* Have received heart or lung transplant
* Receiving mechanical circulatory support
* Patients who have been referred or admitted for Hospice care
* A life expectancy of less than 12 months per physician discretion
* Enrolled in any concurrent study without Boston Scientific written approval
* Devices previously converted to the SRD-1 and withdrawn from the study
* Received a sub-pectoral COGNIS implant prior to February 1, 2011 with a dash number listed in Appendix K of the study protocol
* Known pregnancy or plan to become pregnant within the course of the study
* LV offset is programmed to a value greater than zero

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with CRT-D devices(Heart Failure patients)
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Heart Failure (HF) events | 12 Months
  The primary objectives of this study are to determine how ambulatory sensor measurements change with worsening heart failure, and to develop multisensor detection algorithms. Additional data will be collected to compare sensor measurements against reference measurements when the subject is hospitalized for HF. Data from this study may also be used for determining prospective endpoints and sample sizes for future studies. There are no formal statistical primary or secondary endpoints defined for this study. Therefore, no formal tests of hypothesis will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: John P Boehmer, M.D., Principal Investigator — Milton S Hershey Medical Center, Hershey, Pennsylvania, United States
Locations (99):
- United States (81):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Advanced Arrhythmias, Gilbert, Arizona
  - Baptist Health Medical Center, Little Rock, Arizona
  - Tri-City Cardiology, Mesa, Arizona
  - Cardiovascular Consultants, LTD, Phoenix, Arizona
  - Pima Heart Physicians, PC, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - LAC & USC Medical Center, Los Angeles, California
  - John Muir Medical Center, Oakland, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Daytona Heart Group, Daytona Beach, Florida
  - First Coast Cardiovascular, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Orlando Heart Center, Orlando, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Emory University Hospital, Atlanta, Georgia
  - St Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Wellstar Research Institute, Marietta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - St. Mary's Medical Center, Evansville, Indiana
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Parkview Hospital, Inc., Fort Wayne, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - La Porte Hospital, La Porte, Indiana
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Genesis Medical Center, Davenport, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - St. Joseph Hospital, Lexington, Kentucky
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Providence Hospital, Southfield, Michigan
  - Univeristy of MN Medical Center, Minneapolis, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Bergan Cardiology -Alegent Bergan Mercy Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - Buffalo Cardiology and Pulmonary, Williamsville, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Sanger Heart and Vascular Institution, Charlotte, North Carolina
  - Cardiovascular Research Institute LLC, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Ohio Health Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - St. Elizabeth Health Center, Poland, Ohio
  - Northwest Ohio Cardiology, Toledo, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Rogue Valley Medical Center, Medford, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - The Arrhythmia Institute, Newton, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Cardiovascular Associates of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Inc., Memphis, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - South East Texas Clinical Research, Beaumont, Texas
  - EP Heart, Houston, Texas
  - Heart Hospital of Austin, Houston, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - University of VA Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virgina Commonwealth University Hospital System, Richmond, Virginia
  - Chippenham Medical Center, Richmond, Virginia
  - Monongalia General Hospital, Morgantown, West Virginia
- Faculty Hospital U sv Anny, Brno, Czechia
- University Hospital Jena Cardiology, Jena, Germany
- Prince of Wales Hospital, Shatin, Hong Kong, Hong Kong
- Hungary (3):
  - Hungarian Institute of Cardiology, Budapest
  - Semmelweis University, Cardiovascular Center, Budapest
  - Allami Egeszsegugyi Kozpont (AEK) Hospital, Budapest
- Kaplan Medical Centre, Rehovot, Israel
- Italy (2):
  - Az. Osp. Lancisi, Ancona
  - Ospedale Sacro Cuore Don Calabria, Negrar
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum, Utrecht
- Slovakia (2):
  - The National Institute of Cardiovascular Diseases - NUSCH, Bratislava
  - VUSCH a.s., Košice
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Her Majesty Cardiac Center, Siriraj Hospital, Bangkok
- United Kingdom (2):
  - Golden Jubilee National Hospital, Clydebank
  - The Heart Hospital, London

REFERENCES:
- [Background] J. P. Boehmer, Q. An, Y. Zhang, A. Shih, Variation in daily median respiratory rate identifies patients at higher risk of worsening HF in 30 days, Heart Rhythm, 2013;10(5):S66
- [Background] J. P. Boehmer, Q. An, Y. Zhang, A. Shih, Patients with higher standard deviation in daily median respiratory rate are at higher risk of worsening HF in 30 days, Europace, 2013;15(Suppl 2):ii96
- [Background] J. P. Boehmer, Y. Zhang, K. C. Beck, R. J. Sweeny, Physiologic sensor response to activity level in the MultiSENSE Study, European Journal of Heart Failure, 2013:12 (suppl 1), S194-5
- [Background] J. Hatlestad, S. Mehta, J. Whelan-Schwartz, R. Shankar and J.P. Boehmer, M.D..Night-time Elevation Angles In MultiSENSE Study Are Related To Symptoms of Orthopnea & Paroxysmal Nocturnal Dyspnea, Journal of Cardiac Failure, Vol. 18 No. 8S, Aug 2012, pp. S8
- [Background] J. P. Boehmer, V. Averina, P. Thakur, Y. Zhang, R. J. Sweeny, J. Thompson, Device-based sensors in the MultiSENSE Study: a preliminary view, Journal of Cardiac Failure, Vol. 18 No. 8S, Aug 2012, pp. S18
- [Background] J. P. Boehmer, Y. Zhang, R. J. Sweeny, R. Wariar, Q. An, P. Thakur, V. Averina, J. Thompson, Quantifying circadian variation of multiple physiologic signals in ambulatory heart failure patients, Journal of Cardiac Failure, Vol. 18 No. 8S, Aug 2012, pp. S90
- [Background] J. P. Boehmer, Y. Zhang, K. C. Beck, R. J. Sweeny, Physiologic sensor response to activity level in the MultiSENSE Study, Journal of Cardiac Failure, Vol. 17 No. 8S, Aug 2011, pp. S105
- [Background] J. P. Boehmer, Y. Zhang, R. J. Sweeny, R. Wariar, Q. An, P. Thakur, V. Averina, J. Thompson, Quantifying circadian variation of multiple physiologic signals in ambulatory heart failure patients, European Heart Journal, Vol. 33 Suppl 1, Aug 2012, pp. 162
- [Background] G. Molon, A. Capucci, Y. Zhang, Nicholas Wold, Qi An, Scott Wehrenberg, Existing device diagnostics identify patients at higher risk of worsening heart failure in 30 days, Europace, 2014; 16(Suppl 2):ii123
- [Background] J. Boehmer, Q. An, Y. Zhang, Variation in daily median respiratory rate identifies patients at higher risk of worsening HF in 30 days, Heart & Lung: The Journal of Acute and Critical Care, July 2014; 43(4), pp. 381
- [Background] Michael Cao, Michael Gold, Yi Zhang, Nicholas Wold, Scott Wehrenberg, Qi An, John Boehmer , Implantable device diagnostics identify patients at higher risk of heart failure events in 30 days, Heart & Lung: The Journal of Acute and Critical Care, July 2014; 43(4), pp. 381-2
- [Background] A. Capucci, G. Molon, M R. Gold, Y. Zhang, R. Sweeney, V. Averina, J P. Boehmer, Rapid shallow breathing worsens prior to heart failure decompensation, European Heart Journal, Vol. 35, Suppl 1, Sept. 2014, pp. 678
- [Background] Alessandro Capucci, Giulio Molon, Michael R. Gold, Yi Zhang, Robert Sweeney, Viktoria Averina, John P. Boehmer, Rapid Shallow Breathing Worsens Prior to Heart Failure Decompensation, Journal of Cardiac Failure, Aug. 2014; 20 (8), S14
- [Background] Devi Nair, Roy Gardner, Roy Small, Ramesh Hariharan, Qi An, Pramodsingh H. Thakur, John Boehmer, Baseline S3 Measured using Implanted Accelerometer is more Prominent in Patients with Heart Failure Decompensations, Heart Rhythm, 2015;12(5):S419-420, PO05-45
- [Derived] Capucci A, Wong JA, Gold MR, Boehmer J, Ahmed R, Kwan B, Thakur PH, Zhang Y, Jones PW, Healey JS. Temporal Association of Atrial Fibrillation With Cardiac Implanted Electronic Device Detected Heart Failure Status. JACC Clin Electrophysiol. 2022 Feb;8(2):182-193. doi: 10.1016/j.jacep.2021.09.015. Epub 2021 Nov 24. PMID 35210075
- [Derived] Gardner RS, Thakur P, Hammill EF, Nair DG, Eldadah Z, Stancak B, Ferrick K, Sriratanasathavorn C, Duray GZ, Wariar R, Zhang Y, An Q, Averina V, Boehmer JP. Multiparameter diagnostic sensor measurements during clinically stable periods and worsening heart failure in ambulatory patients. ESC Heart Fail. 2021 Apr;8(2):1571-1581. doi: 10.1002/ehf2.13261. Epub 2021 Feb 22. PMID 33619893
- [Derived] Gardner RS, Singh JP, Stancak B, Nair DG, Cao M, Schulze C, Thakur PH, An Q, Wehrenberg S, Hammill EF, Zhang Y, Boehmer JP. HeartLogic Multisensor Algorithm Identifies Patients During Periods of Significantly Increased Risk of Heart Failure Events: Results From the MultiSENSE Study. Circ Heart Fail. 2018 Jul;11(7):e004669. doi: 10.1161/CIRCHEARTFAILURE.117.004669. PMID 30002113
- [Derived] Boehmer JP, Hariharan R, Devecchi FG, Smith AL, Molon G, Capucci A, An Q, Averina V, Stolen CM, Thakur PH, Thompson JA, Wariar R, Zhang Y, Singh JP. A Multisensor Algorithm Predicts Heart Failure Events in Patients With Implanted Devices: Results From the MultiSENSE Study. JACC Heart Fail. 2017 Mar;5(3):216-225. doi: 10.1016/j.jchf.2016.12.011. PMID 28254128